CLINICAL TRIAL: NCT04207060
Title: Phase 1/2 Trial of Indomethacin in Chronic Pancreatitis (The PAIR Trial)
Brief Title: Trial of Indomethacin in Chronic Pancreatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Santhi Swaroop Vege, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-008193; R21DK117212 (NIH)
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Indomethacin; Endoscopy

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to receive indomethacin or placebo according to a computer generated randomization list composed of randomized blocks of sizes of 2 or 4. Within each block, equal number of subjects will be assigned to indomethacin and placebo. Separate sets of blocks will be provided for Mayo Clinic and Ohio State. The randomization lists will be computer generated by the study statistician (Dr Li), and kept in a secure computer file and paper study binder in the Mayo and Ohio State Research Pharmacies. No investigators or study personnel other than Dr Li will have knowledge of the randomization list. Dr Li will not participate in any aspect of subject recruitment, subject allocation, conduct of the study, or data ascertainment, but will perform data analysis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding: Study medication will be labelled "indomethacin 50 mg or placebo capsule" with the subject's name, hospital or clinic number, study IRB number, and subject number. Placebo and indomethacin capsules will be identical in appearance. The investigators, study coordinator, and clinical caregivers will remain blinded to subject allocation throughout the data ascertainment and data entry phase of the study.
  The success of blinding will be evaluated by asking the investigator, the study coordinator, and the subject the following question during each telephone follow-up visit: "Which treatment group is this subject/were you assigned to: placebo, active drug, or unsure?"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indomethacin (Experimental): The study intervention is oral indomethacin. Indomethacin is an FDA approved, commonly prescribed non-steroidal anti-inflammatory drug (NSAID). Commercially available indomethacin will be utilized in this study. Subjects randomized to the indomethacin arm will take one capsule of 50 mg of Indomethacin orally twice a day for 28 days. Participants will be advised not to make up missed doses. They will be advised to take a dose of study medication on the morning of their follow-up endoscopy, 2 hours prior to their scheduled procedure time, with a sip of water. At the time of follow-up endoscopy they will return any unused study medications.
  Interventions: Drug: Indomethacin; Procedure: Endoscopy for Pancreatic Function Testing
- Placebo (Placebo Comparator): Participants in both study arms will receive study medication, one capsule orally twice a day for 28 days. Those in the placebo arm will take placebo capsules (one capsule) twice a day for a total of 28 days.
  Participants will be advised not to make up missed doses. They will be advised to take a dose of study medication on the morning of their follow-up endoscopy, 2 hours prior to their scheduled procedure time, with a sip of water. At the time of follow-up endoscopy they will return any unused study medication.
  Interventions: Drug: Placebo; Procedure: Endoscopy for Pancreatic Function Testing

INTERVENTIONS:
Drug: Indomethacin — One capsule of 50 mg of indomethacin will be taken orally twice a day for a total of 28 days.
  Arms: Indomethacin
Drug: Placebo — One capsule of lactose not containing active study drug will be taken orally twice a day for a total of 28 days.
  Arms: Placebo
Procedure: Endoscopy for Pancreatic Function Testing — All subjects in the study (regardless of which treatment arm they are randomized to) will undergo an upper endoscopy during which they will receive an endoscopic pancreatic function test. An upper endoscopy will be performed during the baseline visit and at the follow-up visit at day 28 of the treatment (2 endoscopies total per each subject). Specifically, during the upper endoscopy, secretin will be administered intravenously at a weight-based dose of 0.2 mcg/kg over 1 minute. Fluid will be aspirated from the duodenum through the endoscope from 0-10 minutes and 10-20 minutes following secretin administration. The collected fluid will then be sent to the laboratory for analysis.

SUMMARY:
The researchers are trying to find a way to slow down the progression of chronic pancreatitis (CP) and investigate the possibility of the long term treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender, age ≥ 18 years and < 60 years
2. Diagnosed with chronic pancreatitis per American Pancreatic Association guidelines (pancreatic calcifications and/or Cambridge 3-4 changes on CT, MRI, and/or ERCP)
3. Scheduled for an upper GI endoscopic procedure (EGD or EUS) for clinical or research) indications (not conflicting with current investigation).
4. Able to provide written informed consent.
5. Serum creatinine within normal laboratory range, as measured within 30 days of the baseline study endoscopy.
6. For females of reproductive potential: willing to use highly effective contraception while taking study medication and for an additional 5 days after completing study medication.

Exclusion Criteria:

1. Diagnosed with acute pancreatitis requiring hospitalization within the 6 weeks prior to study enrollment.
2. Habitual use of aspirin or non-steroidal anti-inflammatory medications (NSAIDs), defined as use more than once per week.
3. Any use of aspirin or NSAIDs within 1 week of baseline study endoscopy procedure.
4. Allergy to secretin, indomethacin or NSAIDs.
5. History of known chronic renal insufficiency or cirrhosis.
6. History of coronary artery disease, angina pectoris, myocardial infarction, cerebrovascular accident (stroke), or transient ischemic accident (TIA).
7. History of peptic ulcer or gastrointestinal bleeding.
8. Incarcerated.
9. Found to have active GI ulceration at the time of baseline endoscopy.
10. Hospitalized for acute pancreatitis while participating in this research protocol. Participants who are hospitalized for an episode of acute pancreatitis during study participation will be withdrawn from the study, and considered non-accrued.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santhi Vege, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Han S, Vege SS, Hart PA, Saloman JL, Xu J, Li L, Cruz-Monserrate Z, Palermo TM, Hill R, Hao W, Yadav D, Topazian M, Conwell DL. Oral Indomethacin for Chronic Pancreatitis: Results From the PAIR Randomized Placebo-Controlled Trial. Clin Transl Gastroenterol. 2025 Sep 1;16(9):e00888. doi: 10.14309/ctg.0000000000000888. PMID 40622408
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20470484

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants in both study arms will receive study medication, one capsule orally twice a day for 28 days. Those in the placebo arm will take placebo capsules (one capsule) twice a day for a total of 28 days.
  Participants will be advised not to make up missed doses. They will be advised to take a dose of study medication on the morning of their follow-up endoscopy, 2 hours prior to their scheduled procedure time, with a sip of water. At the time of follow-up endoscopy they will return any unused study medication.
  Placebo: One capsule of lactose not containing active study drug will be taken orally twice a day for a total of 28 days.
  Endoscopy for Pancreatic Function Testing: All subjects in the study (regardless of which treatment arm they are randomized to) will undergo an upper endoscopy during which they will receive an endoscopic pancreatic function test. An upper endoscopy will be performed during the baseline visit and at the follow-up visit at day 28 of the treatment (2 endoscopies total per each subject). Specifically, during the upper endoscopy, secretin will be administered intravenously at a weight-based dose of 0.2 mcg/kg over 1 minute. Fluid will be aspirated from the duodenum through the endoscope from 0-10 minutes and 10-20 minutes following secretin administration. The collected fluid will then be sent to the laboratory for analysis.
Period: Overall Study
Arm/Group | Indomethacin | Placebo
Started | 13 | 14
Completed | 11 | 14
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indomethacin | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.6) | 51.1 (11.4) | 53.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Baseline PGE2 Level [Mean (Standard Deviation); unit: pg/ml] | 812.4 (581.4) | 991.6 (1000.3) | 905.3 (790.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Prostaglandin E2 (PGE2) Concentrations
Description: Mean change in PGE2 concentrations in pancreas fluid before and after intervention
Time Frame: Baseline, 28 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 13 | 14
pg/ml | -457.7 (489.8) | -840.4 (865.6)

2. Secondary Outcome: Changes in Pain Interference Score
Description: Measured using the self reported Brief Pain Inventory questionnaire. The pain interference subscale includes 7 items which each utilize a 11-point scale from 0-10, with 10 representing the worst outcome (highest level of pain). The scores from the 7 items are summed to create a total score. Thus, the total score can range from 0-70. The total pain interference score at baseline was then subtracted from the total pain interference score at 28 days to calculate the change in pain interference score.
Time Frame: Baseline, 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 13 | 14
score on a scale | -2.9 (3.6) | -0.4 (1.3)

3. Secondary Outcome: Change in Quality of Life (Mental Health)
Description: Measured using the self reported PROMIS-10 instrument. The PROMIS-10 instrument includes 4 items for mental health, which each have 1-5 scale, with 5 representing the worst outcome. T-scores are then calculated from the raw scores. A mean T-score of 50 represents average health with a standard deviation of 10. Higher scores denote a worse outcome. The mean T-score at baseline was then subtracted from the mean T-score at 28 days to derive the change in mental quality of life..
Time Frame: Baseline, 28 days
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 13 | 14
T-score | -3.8 (10) | 0.1 (6)

4. Secondary Outcome: Change in Pain Composite Score
Description: Assessed using the Brief Pain Inventory (BPI) scale. The pain composite score includes 4 questions from the BPI, each of which is scored on a 0-10 scale with 10 representing the worst outcome (highest level of pain) and 0 representing the best outcome (no pain). The 4 questions assess 1) worst pain, 2) least pain, 3) average pain, and 4) current pain. The mean score of the responses to these 4 questions is calculated to derive the pain composite score. Thus, the pain composite score will also range from 0-10. The mean pain composite score at baseline was then subtracted from the mean pain composite score at 28 days to calculate the change in pain composite score.
Time Frame: Baseline, 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 13 | 14
score on a scale | -1.3 (1.5) | -0.5 (1.4)

5. Secondary Outcome: Change in Quality of Life (Physical Health)
Description: Quality of life measured using the self reported PROMIS-10 instrument. The PROMIS-10 instrument includes 4 items for physical health, which each have a 1-5 scale, with 5 representing the worst outcome. T-scores are then calculated from the raw scores. A T-score of 50 indicates the population mean with a standard deviation of 10. Higher T-scores represent worse outcomes. The mean T-score at baseline was then subtracted from the mean T-score at 28 days to derive the change in physical quality of life.
Time Frame: Baseline, 28 days
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 13 | 14
T-score | 1.6 (5.4) | 1.4 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from initiation of the study intervention to 30 days after completion of the intervention. The follow-up time points were specifically at 7 days, 14 days, 21 days and 58 days following study intervention initiation.
Description: Adverse events and serious adverse events were defined as defined by clinicaltrials.gov
Arm/Group | Indomethacin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 4/13 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin (N=13) | Placebo (N=14)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot Flashes (Endocrine disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include the short treatment period as participants received the study medication for only 28 days, which may be too short to detect a significant biochemical change in a chronic disease such as chronic pancreatitis. Additionally, as this was a Phase 1/2 study, the only dose chosen for the intervention, indomethacin, was 50 mg BID, which may not represent an effective dose to modify chronic pancreatitis. Furthermore, the short follow-up period limits ascertaining long-term effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT04207060/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT04207060/ICF_000.pdf